CLINICAL TRIAL: NCT06983860
Title: Application and Demonstration of Endoscope-assisted Low-temperature Plasma Radiofrequency Ablation Resection of Tonsils
Acronym: A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: People's Hospital of Anshun City of Guizhou Province (Other)
Responsible Party: Principal Investigator, Guangjun Tang, Doctor, People's Hospital of Anshun City of Guizhou Province
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHAnshun1; LC[2025] General 090 (Other Grant/Funding Number: Guizhou Provincial, Department of Science and Technology)
Record Dates: First submitted 2025-04-16; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Tonsil Disease
Keywords: endoscope-assisted; low-temperature plasma; radiofrequency ablation resection; tonsils

STUDY DESIGN:
Intervention Model Description: The prospective study method was adopted, and 100 patients who were admitted to the ward of our hospital for tonsillectomy from January 2025 to December 2025 were recruited as experimental subjects.
  1.1 Main evaluation indicators
  1. Perioperative indexes (operation time, intraoperative blood loss, length of hospital stay) were recorded.
  2. Visual Analogue Scale (VAS): VAS score was performed at 6h, 12h, 24h and 72h after surgery.
  3. Endoscopic examination: On the 2nd, 4th, 2nd and 4th postoperative days, the formation and shedding of tonsillar fossa in the operative area were observed through the mouth under a 70-degree nasal endoscope; Whether there is bleeding or bleeding in the operative area; The recovery of the operative area and the presence or absence of granulation tissue hyperplasia.
  1.2 Secondary evaluation indicators
  1. Postoperative bleeding: Observe and record postoperative bleeding, and calculate the bleeding rate.
  2. The occurrence of complications was recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscope-assisted low-temperature plasma radiofrequency ablation resection of tonsils (Experimental): In this prospective study, 100 patients admitted to our hospital for tonsillectomy from January 2025 to December 2025 will be recruited as experimental subjects. Perioperative indexes (operation time, intraoperative blood loss, length of hospital stay) were recorded. Visual Analogue Scale (VAS) was used: VAS scores were performed at 6h, 12h, 24h and 72h after surgery. Endoscopic examination: On the 2nd, 4th, 2nd and 4th postoperative days, the formation and shedding of tonsillar fossa were observed through the mouth under a 70-degree nasal endoscope. Whether there is bleeding or bleeding in the operative area; The recovery of the operative area and the presence or absence of granulation tissue hyperplasia. Postoperative bleeding and complications were recorded.
  Interventions: Procedure: Application and demonstration of endoscope-assisted low-temperature plasma radiofrequency ablation resection of tonsils

INTERVENTIONS:
Procedure: Application and demonstration of endoscope-assisted low-temperature plasma radiofrequency ablation resection of tonsils — Low temperature plasma radiofofency ablation of tonsil under 70° nasal endoscope can directly view the lesion area on the monitor, clearly enlarge the operating field, and has the advantages of small surgical trauma, good hemostatic effect, light postoperative pain, low probability of postoperative bleeding and quick postoperative recovery of patients, etc. It is a good surgical mode integrating surgery and teaching, and has brought great benefits to patients, and is worth promoting and applying.

SUMMARY:
Low temperature plasma radiofofency ablation of tonsil under 70° nasal endoscope can directly view the lesion area on the monitor, clearly enlarge the operating field, and has the advantages of small surgical trauma, good hemostatic effect, light postoperative pain, low probability of postoperative bleeding and quick postoperative recovery of patients, etc. It is a good surgical mode integrating surgery and teaching, and has brought great benefits to patients, and is worth promoting and applying.

DETAILED DESCRIPTION:
1. Basis for Project Initiation 1.1 Chronic tonsillitis is a common health issue that can significantly impact the patient's quality of life.

Chronic tonsillitis is a common condition in the field of otolaryngology, primarily caused by recurrent episodes of acute tonsillitis that persist and fail to heal, leading to degeneration and necrosis of epithelial cells within the gland. This results in the retention of pathogenic microorganisms and inflammatory exudates, causing blockage of the crypt drainage, which then leads to secondary infections and eventually evolves into chronic inflammation[1]. Clinically, it manifests mainly with symptoms such as frequent colds, discomfort during swallowing, a sensation of something foreign in the throat, dryness in the throat, bad breath, paroxysmal coughing, headaches, and more. In severe cases, it can cause difficulty in breathing, sleep apnea, and even lead to complications like acute nephritis, rheumatic arthritis, heart disease, and scarlet fever, significantly impacting both the physical and mental health of patients, severely affecting their quality of daily life.

1.2 Traditional tonsillectomy is associated with significant trauma and numerous complications, whereas the low-temperature plasma knife causes minimal trauma and offers excellent hemostatic effects.

For chronic tonsillitis patients with recurrent acute tonsillitis, peritonsillar abscess, excessive hypertrophy of tonsils, repeated acute attacks, sleep apnea and neighboring organs involved, surgical treatment is often used in clinic. The surgical methods of tonsillectomy mainly include two categories: one is cold instrument surgery, including traditional tonsillectomy and extrusion; The second is hot instrument surgery, including the application of laser, high-frequency electrotome, low temperature plasma radio frequency surgery. Due to the abundant blood supply of the tonsil, traditional surgery is prone to cause damage and bleeding of arteries and accompanying veins and venous plexus, which affects the surgical field of view and leads to poor hemostatic effect of the wound during the operation, thus prolonging the operation time and affecting the prognosis. Studies have shown that in the process of traditional tonsillectomy, tissues around the knife edge need to be drawn into the sheath, which excessively stretches the tonsils, causing damage to some normal tissues and increasing postoperative pain. In addition, due to insufficient visual field, over-deep resection is likely to result in incomplete intraoperative hemostasis and residual, which is likely to lead to primary postoperative hemorrhage and excessive postoperative pharyngeal activity. It will promote postoperative complications, which is not conducive to postoperative recovery .

With the development of minimally invasive technology, low-temperature plasma radiofrequency ablation has been widely used in various soft tissue surgeries in otorhinolaryngology in recent years, showing advantages such as less trauma, quick postoperative recovery and good prognosis . The application of low-temperature plasma knife in tonsillectomy integrates the functions of surgical cutting, hemostasis and suction, which can clearly separate the tonsil envelope and surrounding tissues, and at the same time draw out blood to clean the wound, thus shortening the operation time and reducing the amount of intraoperative blood loss [15]. The surgical field of view is clear, the damage to the surrounding large blood vessels and muscle tissue is small, and the mechanical damage caused by traditional dissection can be avoided. At the same time, the mucosal tissue of the pharyngeal cavity can be preserved to the maximum extent, which has little impact on the function of the pharyngeal cavity and is conducive to the guarantee of treatment safety. In addition, low-temperature incision wound is more orderly, and can immediately form a protein false film to cover the wound, reduce the stimulation of nerve endings, and help reduce the degree of postoperative pain, so as to promote the early recovery of patients, comprehensively improve the prognosis and improve the quality of life of patients .

The working principle of low-temperature plasma radiofrequency ablation is to use the energy of electric ions to transform the electrolyte between the radiofrequency tool head and the tissue into a plasma layer. The charged ions in the tissue are accelerated by the electric field, and the target tissue cells gradually decompose, atrophy and fall off in the form of molecules. The ablation can be performed under the condition of 40℃ ~ 70℃, and the bleeding can be stopped at the same time. It accurately acts on the inflammation site, greatly improving the accuracy, eliminating the need for compression and sutural hemostasis, making hemostasis more thorough, reducing the probability of primary postoperative bleeding, protecting mucosal integrity, and reducing peripheral vascular and nerve damage. Thus, the occurrence of postoperative bleeding and pharyngeal pain can be reduced, which has a good therapeutic effect in patients with chronic tonsillitis.

Compared with traditional tonsillectomy, low-temperature plasma resection can better preserve tonsil function. Compared with conventional electrotome coagulation, this technique can regulate the radiofrequency energy according to the distance, and the tissue heating is minimal, reducing the risk of deep tissue damage around the tonsil. In recent years, low-temperature plasma resection has been applied more and more widely in the ENT surgical treatment system, and it has been clinically proved that it has achieved relatively ideal effects in reducing postoperative pain and stress reaction and accelerating rehabilitation process.

In summary, low-temperature plasma tonsillectomy for chronic tonsillitis has the advantages of less surgical trauma, less postoperative pain, lower probability of postoperative bleeding, and faster recovery of postoperative patients, which is worthy of clinical promotion and application.

1.3 The endoscopic auxiliary system has the functions of magnification, focusing and high-definition display, which can directly look at the lesion area, making the operation safer.

In recent years, high-definition endoscopic camera system has been applied to tonsillectomy, which has the role of surgical field lighting. By using the endoscopic system, the surgeon can accurately distinguish the pharyngeal mucosa, tonsil envelope, and the fibrous tissue and muscle fiber tissue in the tonsil space. The surgeon can always know the location of the plasma cutter head and the main components of the removed tissue, thus reducing unnecessary intraoperative damage to adjacent tissues, speeding up the surgical process, and reducing the postoperative pain of patients Degree. Compared with the traditional headlamp surgery, it has the advantages of clear operating field, fast intraoperative hemostasis, less damage, light postoperative pain and low bleeding rate, and has a good teaching demonstration effect, which can improve the surgical precision of the surgeon.

Clinical studies have found that most patients with hemorrhage after tonsillar surgery are mainly located in the upper and lower extremum of the tonsillar fossa, because it is impossible to look directly at the lesion under traditional headlamps. After tonsillectomy, the upper tonsillar fossa can be partially exposed, while the lower tonsillar fossa is very difficult to be exposed. These blind areas are the hiding place for hiding bleeding, the tricky place for intraoperative hemostasis and the high incidence of postoperative bleeding. It has been reported that the incidence of hemorrhage after tonsillectomy is 5.9% ~ 13.9% in foreign countries. The incidence in China ranges from 2% to 8%, with an average of 3%. Excessive blood loss can lead to anemia and hemorrhagic shock in patients, even life-threatening, which brings great pain and mental pressure to patients and their families, as well as prolongation of hospital stay and increased medical costs.

With the assistance of 70° nasal endoscopy, any area of the operation can be observed in an all-round field of vision without dead Angle, and can be displayed in high-definition on the display screen, which helps to find hidden bleeding and exposed blood vessels in the upper and lower poles of the tonsil fossa that cannot be detected under direct vision, and precisely hemostasis of the bleeding site, which not only reduces unnecessary damage to adjacent tissues caused by blind electrocoagulation, but also reduces the postoperative pain of patients Thus, the intraoperative hemostasis time is shortened and the incidence of postoperative bleeding is reduced. It has brought some benefits to patients and medical staff, and has a good application prospect and popularization role.

In summary, low-temperature plasma radiofofency ablation of tonsil under 70° nasal endoscope can directly view the lesion area on the monitor, clearly enlarge the operating field, and has the advantages of small surgical trauma, good hemostasis, light postoperative pain, low probability of postoperative bleeding, and quick postoperative recovery of patients, etc. It is a good surgical mode integrating surgery and teaching, and has brought great benefits to patients. It is worth promoting and applying.

At present, many large hospitals at home and abroad have gradually carried out endoscopic low-temperature plasma ablation of tonsils. In view of the difficulty in controlling the endoscopic tonsil resection and endoscopic hemostasis, hospitals in our province and local areas rarely carry out endoscopic low-temperature plasma radiofofency ablation in inpatients since 2023. It has been fully certified and affirmed in some patients, but due to the small sample size, it cannot be better promoted and applied. Therefore, this study intends to increase publicity through this project, form standardized diagnosis and treatment technology schemes and surgical procedures, and encourage more doctors to choose this operation for patients, so as to reduce complications and improve patients' medical experience. Enhance the recognition of regional medical level, thereby indirectly increasing the economic benefit level of hospitals and departments, and reducing the economic burden of patients.

ELIGIBILITY:
Inclusion Criteria:

1. History of recurrent acute attacks of chronic tonsillitis, with the number of attacks >3 times per year for more than 2 years;
2. accompanied by snoring, choking and apnea during night sleep;
3. Age 3-65 years old, gender is not limited;
4. No major systemic diseases, such as cardiovascular and cerebrovascular diseases, liver and kidney insufficiency, hematopoietic system diseases;
5. Subjects who can understand and abide by the research procedures and voluntarily participate in the experiment by signing the informed consent form (the informed consent is signed by themselves or their legal representatives).

Exclusion Criteria:

1. cardiopulmonary insufficiency;
2. Patients with systemic blood diseases;
3. Patients with acute and chronic bronchial or lung infections;
4. Complicated with severe cardiovascular system disease or hepatic and renal insufficiency;

6) Patients with mental abnormalities or who do not cooperate with treatment 7) Researchers who are participating in other trials.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative indexes | intraoperative
  operation time, intraoperative blood loss, length of hospital stay
Visual Analogue Scale (VAS) | VAS score was performed at 6h, 12h, 24h and 72h after surgery
  VAS score is a widely used subjective assessment method for pain assessment. Using a walking scale about 10cm long, one side is marked with 10 scales, and the two ends are respectively "0" and "10". 0 indicates no pain, and 10 indicates unbearable pain. The patient is asked to mark the pain value and record it.
Endoscopic examination | On the 2nd, 4th, 2nd and 4th postoperative days
  the formation and shedding of tonsillar fossa in the operative area were observed through the mouth under a 70-degree nasal endoscope; Whether there is bleeding or bleeding in the operative area; The recovery of the operative area and the presence or absence of granulation tissue hyperplasia

SECONDARY OUTCOMES:
Postoperative bleeding | Within 1 month after surgery
  Observe and record postoperative bleeding, and calculate the bleeding rate.
The occurrence of complications was recorded. | Within 1 month after surgery
  Were there any complications within 1 month after surgery and what were the complications

CONTACTS AND LOCATIONS:
Overall Officials: Jun G Tang, Dr, Study Chair — principal

IPD SHARING:
Plan to Share IPD: Yes
The data will be published online as a paper
Supporting Information: Study Protocol
Time Frame: December 2025 to December 2026
Access Criteria: The data and content of my published study can be accessed by email or downloaded online